CLINICAL TRIAL: NCT00035737
Title: Vascular Function in the Framingham Third Generation
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1050; R01HL070100 (NIH)
Record Dates: First submitted 2002-05-04; First posted 2002-05-06 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To investigate the role of endothelial dysfunction and increased vascular stiffness as contributors to the pathogenesis of cardiovascular disease.

DETAILED DESCRIPTION:
BACKGROUND:

Increasingly, researchers understand that endothelial dysfunction and increased vascular stiffness contribute to the pathogenesis of cardiovascular disease (CVD). The Framingham Heart Study (FHS) has been examining vascular function in about 3600 middle-aged and elderly participants of the FHS Offspring and minority OMNI cohorts.

DESIGN NARRATIVE:

The study characterizes vascular function by performing noninvasive studies of endothelial function with brachial ultrasound flow-mediated dilation, and of vascular stiffness with arterial tonometry, in 3850 adult offspring of the FHS Offspring and OMNI cohorts. The total of over 7000 vascular examinations in an extensively studied multi-generational community-based cohort provides the opportunity to characterize the environmental and genetic determinants, and the prognosis of altered vascular function. The study hypotheses are: vascular function is determined by both environmental and genetic factors; endothelial function and vascular stiffness phenotypes are associated with each other: and vascular dysfunction predisposes to the development of hypertension (HTN) and cardiovascular disease.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-05; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emelia Benjamin — Boston University

REFERENCES:
- [Background] Vita JA, Keaney JF Jr, Larson MG, Keyes MJ, Massaro JM, Lipinska I, Lehman BT, Fan S, Osypiuk E, Wilson PW, Vasan RS, Mitchell GF, Benjamin EJ. Brachial artery vasodilator function and systemic inflammation in the Framingham Offspring Study. Circulation. 2004 Dec 7;110(23):3604-9. doi: 10.1161/01.CIR.0000148821.97162.5E. Epub 2004 Nov 29. PMID 15569842
- [Background] Benjamin EJ, Larson MG, Keyes MJ, Mitchell GF, Vasan RS, Keaney JF Jr, Lehman BT, Fan S, Osypiuk E, Vita JA. Clinical correlates and heritability of flow-mediated dilation in the community: the Framingham Heart Study. Circulation. 2004 Feb 10;109(5):613-9. doi: 10.1161/01.CIR.0000112565.60887.1E. PMID 14769683
- [Background] Vita JA. Endothelial function and clinical outcome. Heart. 2005 Oct;91(10):1278-9. doi: 10.1136/hrt.2005.061333. No abstract available. PMID 16162617
- [Background] Vita JA, Mitchell GF. Effects of shear stress and flow pulsatility on endothelial function: insights gleaned from external counterpulsation therapy. J Am Coll Cardiol. 2003 Dec 17;42(12):2096-8. doi: 10.1016/j.jacc.2003.09.020. No abstract available. PMID 14680733
- [Background] Ganz P, Vita JA. Testing endothelial vasomotor function: nitric oxide, a multipotent molecule. Circulation. 2003 Oct 28;108(17):2049-53. doi: 10.1161/01.CIR.0000089507.19675.F9. No abstract available. PMID 14581383